CLINICAL TRIAL: NCT06156722
Title: The Combination of Sperm Selection by IMSI and Hyaluronic Acid Binding Assay Improves ICSI Outcomes: A Randomized Prospective Sibling-oocytes Study
Brief Title: The Combination of Sperm Selection by IMSI and Hyaluronic Acid Binding Assay May Improve ICSI Outcome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Assuta Medical Center (Other); Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yael Yagur, Consultant, Obstetrics and Gynaecology Department. Principal investigator. Lecturer., Meir Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MEIRIMSIRCT
Record Dates: First submitted 2023-11-02; First posted 2023-12-05 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Fertility Issues
Keywords: IMSI; SpermSlow; Sperm selection; ICSI outcome; Sibling-oocytes study
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The IMSI-only group (Active Comparator): The IMSI-only group
  Interventions: Procedure: Sperm selection by IMSI
- IMSI with SpermSlow group (Active Comparator): IMSI with SpermSlow group
  Interventions: Procedure: Sperm selection by IMSI and spermslow
- Mixed embryo group (No Intervention): Mixed embryo group

INTERVENTIONS:
Procedure: Sperm selection by IMSI — Intracytoplasmic morphologically selected sperm injection (IMSI) is a sperm selection method used in intracytoplasmic sperm injection (ICSI)
  Arms: The IMSI-only group
Procedure: Sperm selection by IMSI and spermslow — Intracytoplasmic morphologically selected sperm injection (IMSI) is a sperm selection method used in intracytoplasmic sperm injection (ICSI) + spermslow
  Arms: IMSI with SpermSlow group

SUMMARY:
In this prospective randomized sibling-oocytes blinded study, investigators examine the combination of two sperm selection methods that logically seem to complete each other, and potentially may improve ICSI outcomes.

The methods include the selection of the optimal spermatozoa based on its morphology by IMSI, together with its physiological function of binding to HA by Spermslow (SS).

The current study compared a group of ET after sperm selection by IMSI with SS to a group of ET after sperm selection by IMSI-only without SS, and to a mixed ET group where two embryos were transferred, one after IMSI-only and the other one after IMSI with SS.

ELIGIBILITY:
Inclusion Criteria:

females ages 38 or younger retrieval of at least 5 mature oocytes and fresh ejaculate samples

Exclusion Criteria:

frozen embryos surgically extracted sperm preparations embryo-biopsy cycles

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Based on sperm and ovum during IVF procedure
Enrollment: 189 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Pregnancy and delivery rates | Within up to 10 month from treatment
  Pregnancy and delivery rates

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel